CLINICAL TRIAL: NCT01077076
Title: Randomized, Placebo-Controlled, Crossover Pharmacodynamic Study Comparing the Effects of Two Different Forms of Omeprazole
Brief Title: Pharmacodynamic Study Comparing the Effects of Two Different Forms of Omeprazole (P07812) (COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 18132; P07812 (Other: Merck)
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Results first posted 2010-04-02 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Intragastric Acidity
Keywords: Gastric Acid; Human Experimentation
MeSH Terms: interventions — omeprazole, sodium bicarbonate drug combination; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Zegerid OTC Capsules (Experimental): 20 mg omeprazole and 1100 mg sodium bicarbonate
  Interventions: Drug: Zegerid
- Prilosec OTC™ tablets containing 20 mg-equivalent omeprazole (Active Comparator): 20.6 mg omeprazole-magnesium complex.
  Interventions: Drug: Prilosec OTC™ Tablets
- Placebo (Placebo Comparator): Inert substance
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Zegerid — Zegerid taken once daily for 11 days.
  Arms: Zegerid OTC Capsules
Drug: Prilosec OTC™ Tablets — Prilosec OTC™ Tablets taken once daily for 11 days.
  Arms: Prilosec OTC™ tablets containing 20 mg-equivalent omeprazole
Other: Placebo — Placebo taken once daily for 11 days.
  Arms: Placebo

SUMMARY:
This randomized, crossover study is to evaluate the early effectiveness, defined as effect on intragastric pH during the first 4 hours after dosing, of Zegerid, Prilosec over-the-counter (OTC) Tablets, and placebo on the 4th day of treatment to inhibit acid secretion. Additional purposes are to:

1. provide pharmacodynamic evidence comparing 24-hr inhibition of acid secretion on the 1st, 4th, and 11th days of dosing with each of the indicated treatments;
2. compare Zegerid and Prilosec OTC for achieving their steady-state effects for controlling 24-hr gastric acidity at steady-state on the 4th and 11th day of dosing.
3. evaluate early effectiveness, defined as effect on intragastric pH during the first 4 hours after administration, of Zegerid, Prilosec OTC Tablets, and placebo on acid inhibition at steady-state when administered on the 11th day of dosing.

DETAILED DESCRIPTION:
Participants were randomized in a 3-way crossover design and received, in random order, Zegerid OTC Capsules (20 mg omeprazole and 1100 mg sodium bicarbonate), Prilosec OTC Tablets (20 mg-equivalent omeprazole), and Placebo Capsules. Participants received each treatment for 11 days. There was a minimum of a 2-week washout period between treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-lactating, non-pregnant female subjects who are 18-65 years of age.
* Physical examination findings within normal limits for age.

Exclusion Criteria:

* History of hypersensitivity, allergy or intolerance to omeprazole, or other proton pump inhibitors
* History of peptic ulcer disease or other acid related gastrointestinal symptoms or heartburn with a frequency of more than one/month.
* Participation in any study of an investigational treatment in the 30 Days before Screening or participation in another study at any time during the period of this study
* Any significant medical illness that would contraindicate participation in the study
* Gastrointestinal disorder or surgery leading to impaired drug absorption
* Any abnormal Screening laboratory value that is clinically significant in the investigator's opinion
* Current use of any prescription or OTC medications that affect gastrointestinal function.
* Currently using or having a history of frequent use of antacids, OTC or prescription (Rx) histamine-2 (H2) receptor antagonists, or OTC or Rx use of proton pump inhibitors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Zegerid/Prilosec/Placebo: Participants received Zegerid over-the-counter (OTC) Capsules (20 mg omeprazole and 1100 mg sodium bicarbonate) in the first intervention, Prilosec OTC Tablets (20 mg-equivalent omeprazole) in the second intervention (after the washout period), and Placebo Capsules in the third intervention (after the washout period).
- Zegerid/Placebo/Prilosec: Participants received Zegerid OTC Capsules (20 mg omeprazole and 1100 mg sodium bicarbonate) in the first intervention, Placebo Capsules in the second intervention (after the washout period), and Prilosec OTC Tablets (20 mg-equivalent omeprazole) in the third intervention (after the washout period).
- Prilosec/Zegerid/Placebo: Participants received Prilosec OTC Tablets (20 mg-equivalent omeprazole) in the first intervention, Zegerid OTC Capsules (20 mg omeprazole and 1100 mg sodium bicarbonate) in the second intervention (after the washout period), and Placebo Capsules in the third intervention (after the washout period).
- Prilosec/Placebo/Zegerid: Participants received Prilosec OTC Tablets (20 mg-equivalent omeprazole) in the first intervention, Placebo Capsules in the second intervention (after the washout period), and Zegerid OTC Capsules (20 mg omeprazole and 1100 mg sodium bicarbonate) in the third intervention (after the washout period).
- Placebo/Zegerid/Prilosec: Participants received Placebo Capsules in the first intervention, Zegerid OTC Capsules (20 mg omeprazole and 1100 mg sodium bicarbonate) in the second intervention (after the washout period), and Prilosec OTC Tablets (20 mg-equivalent omeprazole) in the third intervention (after the washout period).
- Placebo/Prilosec/Zegerid: Participants received Placebo Capsules in the first intervention, Prilosec OTC Tablets (20 mg-equivalent omeprazole) in the second intervention (after the washout period), and Zegerid OTC Capsules (20 mg omeprazole and 1100 mg sodium bicarbonate) in the third intervention (after the washout period).
Period: First Intervention
Arm/Group | Zegerid/Prilosec/Placebo | Zegerid/Placebo/Prilosec | Prilosec/Zegerid/Placebo | Prilosec/Placebo/Zegerid | Placebo/Zegerid/Prilosec | Placebo/Prilosec/Zegerid
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5 | 5 | 5
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: Washout Period of 2 Weeks
Arm/Group | Zegerid/Prilosec/Placebo | Zegerid/Placebo/Prilosec | Prilosec/Zegerid/Placebo | Prilosec/Placebo/Zegerid | Placebo/Zegerid/Prilosec | Placebo/Prilosec/Zegerid
Started | 4 | 5 | 5 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Zegerid/Prilosec/Placebo | Zegerid/Placebo/Prilosec | Prilosec/Zegerid/Placebo | Prilosec/Placebo/Zegerid | Placebo/Zegerid/Prilosec | Placebo/Prilosec/Zegerid
Started | 4 | 5 | 5 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period of 2 Weeks
Arm/Group | Zegerid/Prilosec/Placebo | Zegerid/Placebo/Prilosec | Prilosec/Zegerid/Placebo | Prilosec/Placebo/Zegerid | Placebo/Zegerid/Prilosec | Placebo/Prilosec/Zegerid
Started | 4 | 5 | 5 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Zegerid/Prilosec/Placebo | Zegerid/Placebo/Prilosec | Prilosec/Zegerid/Placebo | Prilosec/Placebo/Zegerid | Placebo/Zegerid/Prilosec | Placebo/Prilosec/Zegerid
Started | 4 | 5 | 5 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death in the participant's family | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (7.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Percent Time With Intragastric pH>4 During the First 4 Hours Following Administration on Day 4 of Treatment
Description: Early effectiveness of treatment is evaluated as the percent time with intragastric pH>4 during the first 4 hours following administration of respective treatments
Time Frame: 4 hours after dose on Day 4
Population: Pharmacodynamic-Evaluable Population: All participants who presented valid data from all three study periods.
  One participant was dropped from the Pharmacodynamic-Evaluable Population in the Prilosec OTC Tablets group because of invalid pH tracings at Day 4. Therefore, the number of participants included at Day 4 in this group was 26.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Groups:
- Prilosec OTC Tablets: 20 mg-equivalent omeprazole
Arm/Group | Zegerid OTC Capsules | Prilosec OTC Tablets | Placebo Capsules
Number analyzed (Participants) | 27 | 27 | 27
Percentage of Time | 53.265 (27.588) | 46.933 (21.885) | 17.215 (15.432)

ADVERSE EVENTS:
Arm/Group | Zegerid OTC Capsules | Prilosec OTC Tablets | Placebo Capsules
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 2/30 | 2/29 | 0/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zegerid OTC Capsules (N=30) | Prilosec OTC Tablets (N=29) | Placebo Capsules (N=29)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Schering-Plough HealthCare Products, Inc. reserves all publication and presentation rights.